CLINICAL TRIAL: NCT05674929
Title: An Open-Label, Phase 2a Single Dose Study in Patients With Alcohol Use Disorder
Brief Title: An Open-Label, Single Dose Study in Patients With Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beckley Psytech Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-003-203
Record Dates: First submitted 2022-12-13; First posted 2023-01-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BPL-003 arm (Experimental)
  Interventions: Drug: BPL-003

INTERVENTIONS:
Drug: BPL-003 — A single dose administered intranasally

SUMMARY:
An open-label, Phase 2a study to evaluate the safety, tolerability, and pharmacodynamic effects of a single intranasal dose of BPL-003 combined with relapse prevention psychological support, to explore the potential effects on alcohol use and related symptoms in patients with Alcohol Use Disorder.

DETAILED DESCRIPTION:
Approximately 12 eligible participants will be receive a single dose of BPL-003, given intranasally, with 12 weeks of follow-up assessments. Psychological support will be given before, during and after dosing

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Age 18 to 64 years at Screening.
3. Diagnosed with moderate to severe AUD.
4. Minimum of 4 heavy drinking days in the 28 days before Screening.
5. No more than 14 days have elapsed since the last HDD or completion of detoxification, with no HDD in the 72 hours prior to dosing and no alcohol at all in the 24 hours prior to dosing
6. Willing to abstain from using recreational drugs from Screening until end of the study
7. Willing to abstain from smoking during their time in the clinic on the day of dosing.
8. Willing to refrain from psychedelic drug use from Screening until the end of the study.
9. Living in stable/secure accommodation in the community.
10. In possession of a personal mobile phone and able to nominate at least one locator individual (eg, a family member, friend, or recovery mentor), with a verifiable address and a telephone number to assist with the arrangement of follow-up appointments.

Exclusion Criteria:

1. Personal or first-degree family history of schizophrenia, bipolar disorder, psychotic disorder, delusional disorder, paranoid disorder or schizoaffective disorder.
2. Any major psychiatric disorders, with the exception of mild or moderate anxiety and/or depression.
3. A clinical diagnosis of post-traumatic stress disorder.
4. Suicide ideation or behaviour or self-injurious behaviours within the 12 months before screening
5. Regular use of or dependence on other drugs other than caffeine or nicotine.
6. Any self-reported use of psychedelic compounds in the past 6 months.
7. History of seizures.
8. Patients who are exhibiting any signs of alcohol withdrawal on dosing day.
9. Positive for alcohol on dosing day.
10. Positive urine drug screen for illicit drugs or drugs of abuse.
11. Any nasal obstruction, blockage, or symptoms of congestion.
12. Any personal or family history of malignant hyperthermia.
13. Patients with an uncontrolled cardiovascular disorder that, in the opinion of the Investigator, may interfere with the interpretation of study results or constitute a health risk for the patient if he/she takes part in the study.
14. Uncontrolled or insulin-dependent diabetes.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with treatment emergent adverse events | Up to12 weeks
Percentage of patients with clinically significant abnormal laboratory tests | Up to12 weeks
Percentage of patients with clinically significant abnormal vital signs | Up to12 weeks
Percentage of patients with suicidal ideation and changes in Columbia Suicidality Rating Scores (CSSRS) | Up to12 weeks
Readiness for discharge questionnaire | 1 Day
Reactivation Questionnaire | Up to 12 weeks
  Measure the frequency, emotional valence and functional impact of any re-activation events in the study

SECONDARY OUTCOMES:
Effects on the Mystical Experience Questionnaire (MEQ30) | 1 Day
Effects on the Ego Dissolution Inventory (EDI) | 1 Day
Percentage of patients experiencing a complete mystical experience, as assessed by the Mystical Experience Questionnaire (MEQ30) | 1 Day
Percentage of patients experiencing a an ego dissolution, as assessed by the Ego Dissolution Inventory (EDI) | 1 Day
Description of the BPL-003 subjective experience data, from a qualitative interview | 1 Day
Feedback from therapists on the frequency and duration of psychotherapy sessions, therapy manual and overall therapy model | 1 Day

OTHER OUTCOMES:
Timeline Follow-Back (TLFB) interview to assess the Percentage of Abstinent days (PAD) in 85d prior D-3 (or start of detox) vs PAD on d14, d28, d56, d84 (with biomarker verification). | Up to 12 weeks
Timeline Follow-Back (TLFB) interview to assess Percentage of Heavy Drinking Days (PHDD) in 85d prior D-3 (or start of detox) vs PHDD post-dosing measured on d14, d28, d56, d84 | Up to 12 weeks
Timeline Follow-Back (TLFB) interview to assess Percentage of Drinking Days (PDD) in 85d prior D-3 (or start of detox) vs PDD post-dosing measured on d14, d28, d56, d84 | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: VP & Head of Clinical Development, PhD, Study Director — Beckley Psytech Ltd
Locations (2):
- United Kingdom (2):
  - Clerkenwell Health, London
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No
Due to the UK GDPR, individual participant data will not be shared publicly. Group data will be presented in publication after study completion.